CLINICAL TRIAL: NCT03822325
Title: Inflammatory Mediators as Potential Non-Invasive Biomarkers and Understanding the Mechanism of Remodeling in Tissue Biopsies in Subjects With Eosinophilic Esophagitis: A Pilot Study
Brief Title: Inflammatory Mediators as Potential Non-Invasive Biomarkers in Subjects With Eosinophilic Esophagitis
Status: Active, not recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Joshua Wechsler, Attending Physician, Gastroenterology, Hepatology & Nutrition, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2010-14155
Record Dates: First submitted 2018-08-16; First posted 2019-01-30 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — The investigators collected biopsies, blood, and urine from enrolled participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort

SUMMARY:
The investigators seek to assess esophageal inflammation or lack of it in response to treatment with a novel non-invasive method that would measure eosinophil-associated inflammatory mediators in the blood and urine to determine the presence of active Eosinophilic Esophagitis. For these purposes, the investigators will correlate esophageal inflammatory mediators measured in blood and urine with histological findings identified on esophageal mucosal biopsies. Additionally, biopsies associated mediators will be assessed relative to clinical phenotype and outcome.

DETAILED DESCRIPTION:
The diagnosis, assessment of recurrence of inflammation, response to treatment and remission in EoE are all currently based on histological evaluation of upper endoscopic pinch esophageal biopsies. Obtaining biopsies for histological evaluation by this procedure is both invasive and expensive. The purpose of our longitudinal prospective study is to evaluate and quantify a panel of novel non-invasive eosinophilic inflammatory biomarkers in the blood and urine of subjects with EoE and compare their presence and levels with the presence or absence of measures of inflammation in esophageal biopsies. While evaluation of esophageal biopsies with 15 or more eosinophils per high power field is the gold standard for diagnosis of EoE, novel predictors of clinical outcome remain unclear. The objective is to identify one or more sensitive and specific non-invasive biomarkers that could be used to monitor esophageal inflammation, and identify novel tissue-based markers that identify phenotype and outcome. This would eliminate the need for invasive serial surveillance endoscopies for the purpose of evaluating for recurrence of inflammation or response to standard therapy since symptoms alone do not adequately correlate with either the presence or absence of disease activity (inflammation) in the esophagus of patients with EoE.

ELIGIBILITY:
Inclusion Criteria:

* Patient ages 1-18 undergoing upper endoscopy for suspected esophageal disease or esophageal inflammation or has histologically confirmed esophageal inflammation may be included in this study

Exclusion Criteria:

* Patients with a history or current diagnosis of esophageal malignancy or subjects with graft versus host disease will be excluded from the study.
* Patients that are considered at high risk for biopsies at the discretion of the child's physician and/or the researcher
* Patients with known bleeding disorders or patients with illnesses where bleeding would pose a threat to their health
* Diagnosis other than Eosinophilic Esophagitis (EoE) i.e. Inflammatory Bowel Disease (IBD), Gastroesophageal Reflux Disease (GERD)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Any patient undergoing a clinically indicated upper endoscopy with biopsy for suspected esophageal inflammation or esophageal disease, or who has histologically confirmed esophageal inflammation may be asked to enroll in this study. The investigators plan to recruit subjects for two years, and enroll up to 150 patients. The patients with a confirmed diagnosis of EoE will be followed in the study for two years after enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Correlate RNA and protein measures from esophageal biopsies with histologic, endoscopic and clinical aspects of disease along with non-invasive biomarkers | 5 years
  Frozen biopsies and archived slides from EoE patients and controls will be used in testing molecules released by or expressed on the cell surface of inflammatory cells. The molecules will be assessed using RNA sequencing, ELISA, and immunohistochemistry. This information will be correlated with eosinophil counts along with endoscopy findings, treatment outcomes and clinical measures of the disease such as symptoms, atopic co-morbidities, and demographics.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Wechsler, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Barry Wershil, MD, Principal Investigator — Ann & Robert H. Lurie Children's Hospital fo Chicago
Locations (2):
- United States (2):
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Illinois at Chicago (UIC), Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dellon ES, Hirano I. Epidemiology and Natural History of Eosinophilic Esophagitis. Gastroenterology. 2018 Jan;154(2):319-332.e3. doi: 10.1053/j.gastro.2017.06.067. Epub 2017 Aug 1. PMID 28774845
- [Background] O'Shea KM, Aceves SS, Dellon ES, Gupta SK, Spergel JM, Furuta GT, Rothenberg ME. Pathophysiology of Eosinophilic Esophagitis. Gastroenterology. 2018 Jan;154(2):333-345. doi: 10.1053/j.gastro.2017.06.065. Epub 2017 Jul 27. PMID 28757265
- [Background] Jensen ET, Kappelman MD, Martin CF, Dellon ES. Health-care utilization, costs, and the burden of disease related to eosinophilic esophagitis in the United States. Am J Gastroenterol. 2015 May;110(5):626-32. doi: 10.1038/ajg.2014.316. Epub 2014 Sep 30. PMID 25267327
- [Background] Furuta GT, Katzka DA. Eosinophilic Esophagitis. N Engl J Med. 2015 Oct 22;373(17):1640-8. doi: 10.1056/NEJMra1502863. PMID 26488694
- [Background] Steinbach EC, Hernandez M, Dellon ES. Eosinophilic Esophagitis and the Eosinophilic Gastrointestinal Diseases: Approach to Diagnosis and Management. J Allergy Clin Immunol Pract. 2018 Sep-Oct;6(5):1483-1495. doi: 10.1016/j.jaip.2018.06.012. Epub 2018 Jul 3. PMID 30201096
- [Background] Dellon ES, Liacouras CA, Molina-Infante J, Furuta GT, Spergel JM, Zevit N, Spechler SJ, Attwood SE, Straumann A, Aceves SS, Alexander JA, Atkins D, Arva NC, Blanchard C, Bonis PA, Book WM, Capocelli KE, Chehade M, Cheng E, Collins MH, Davis CM, Dias JA, Di Lorenzo C, Dohil R, Dupont C, Falk GW, Ferreira CT, Fox A, Gonsalves NP, Gupta SK, Katzka DA, Kinoshita Y, Menard-Katcher C, Kodroff E, Metz DC, Miehlke S, Muir AB, Mukkada VA, Murch S, Nurko S, Ohtsuka Y, Orel R, Papadopoulou A, Peterson KA, Philpott H, Putnam PE, Richter JE, Rosen R, Rothenberg ME, Schoepfer A, Scott MM, Shah N, Sheikh J, Souza RF, Strobel MJ, Talley NJ, Vaezi MF, Vandenplas Y, Vieira MC, Walker MM, Wechsler JB, Wershil BK, Wen T, Yang GY, Hirano I, Bredenoord AJ. Updated International Consensus Diagnostic Criteria for Eosinophilic Esophagitis: Proceedings of the AGREE Conference. Gastroenterology. 2018 Oct;155(4):1022-1033.e10. doi: 10.1053/j.gastro.2018.07.009. Epub 2018 Sep 6. PMID 30009819
- [Background] Godwin B, Wilkins B, Muir AB. EoE disease monitoring: Where we are and where we are going. Ann Allergy Asthma Immunol. 2020 Mar;124(3):240-247. doi: 10.1016/j.anai.2019.12.004. Epub 2019 Dec 9. PMID 31830586
- [Background] Carlson DA, Lin Z, Hirano I, Gonsalves N, Zalewski A, Pandolfino JE. Evaluation of esophageal distensibility in eosinophilic esophagitis: an update and comparison of functional lumen imaging probe analytic methods. Neurogastroenterol Motil. 2016 Dec;28(12):1844-1853. doi: 10.1111/nmo.12888. Epub 2016 Jun 16. PMID 27311807
- [Background] Abonia JP, Wen T, Stucke EM, Grotjan T, Griffith MS, Kemme KA, Collins MH, Putnam PE, Franciosi JP, von Tiehl KF, Tinkle BT, Marsolo KA, Martin LJ, Ware SM, Rothenberg ME. High prevalence of eosinophilic esophagitis in patients with inherited connective tissue disorders. J Allergy Clin Immunol. 2013 Aug;132(2):378-86. doi: 10.1016/j.jaci.2013.02.030. Epub 2013 Apr 19. PMID 23608731
- [Background] Tinkle BT, Levy HP. Symptomatic Joint Hypermobility: The Hypermobile Type of Ehlers-Danlos Syndrome and the Hypermobility Spectrum Disorders. Med Clin North Am. 2019 Nov;103(6):1021-1033. doi: 10.1016/j.mcna.2019.08.002. PMID 31582002
- [Background] Huang KZ, Dellon ES. Increased prevalence of autonomic dysfunction due to postural orthostatic tachycardia syndrome in patients with eosinophilic gastrointestinal disorders. J Gastrointestin Liver Dis. 2019 Mar;28(1):47-51. doi: 10.15403/jgld.2014.1121.281.syd. PMID 30851172
- [Background] Fikree A, Aziz Q, Sifrim D. Mechanisms underlying reflux symptoms and dysphagia in patients with joint hypermobility syndrome, with and without postural tachycardia syndrome. Neurogastroenterol Motil. 2017 Jun;29(6). doi: 10.1111/nmo.13029. Epub 2017 Feb 12. PMID 28191707